CLINICAL TRIAL: NCT04669704
Title: Clinical and Economic Effectiveness of a Tele-rehabilitation Evidence-based Tablet Application for Rehabilitation in Traumatic Bone and Soft Injuries of the Hand, Wrist and Fingers.
Brief Title: Effectiveness of a Tele-Rehabilitation Evidence-based Tablet App for Rehabilitation in Traumatic Bone and Soft Injuries of the Hand, Wrist and Fingers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Maria Dolores Cortes Vega, PhD Professor, University of Seville, University of Seville
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIN-0143-2017
Record Dates: First submitted 2020-11-22; First posted 2020-12-17 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Soft Tissue Injuries; Distal Radius Fracture; Metacarpal Fracture; Carpal Fracture; Carpal Tunnel Syndrome; Thumb Osteoarthritis; Dupuytren's Disease
MeSH Terms: conditions — Soft Tissue Injuries; Wrist Fractures; Carpal Tunnel Syndrome; Dupuytren Contracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet application (Experimental): A protocol of exercises based on the current scientific evidence will be provided through a tablet application. A follow-up of the use of the application will be carried out. A minimum of 4-week home exercise intervention will be performed, which will have to be carried out daily by the patient autonomously at home for at least 5 days per week, starting after baseline measurement.
  The exercise program will be individualized according to each pathology.
  Interventions: Other: Experimental: Tablet application
- Conventional treatment (Active Comparator): In the control condition, participants will receive a home exercise program on paper. The exercise program will be the conventionally prescribed one by the Andalusian Public Health Service. Participants will be told to perform exercises during a minimum of 4 week at home for at least 5 days per week, starting after baseline measurement.
  Interventions: Other: Comparator: Conventional treatment

INTERVENTIONS:
Other: Experimental: Tablet application — A protocol of exercises based on the current scientific evidence will be provided through a tablet application. A follow-up of the use of the application will be carried out. A minimum of 4-week home exercise intervention will be performed, which will have to be carried out daily by the patient autonomously at home for at least 5 days per week, starting after baseline measurement.
  The exercise program will be individualized according to each pathology.
  Arms: Tablet application
Other: Comparator: Conventional treatment — In the control condition, participants will receive a home exercise program on paper. The exercise program will be the conventionally prescribed one by the Andalusian Public Health Service. Participants will be told to perform exercises during a minimum of 4 week at home for at least 5 days per week, starting after baseline measurement.
  Arms: Conventional treatment

SUMMARY:
Trauma and soft injuries of the wrist, hand and fingers have a high incidence, and large social and healthcare costs are generated, mainly due to productivity loss. Therapeutic exercises must be part of the treatment and in the last 10 years the scientific literature highlights the need for the inclusion of the sensorimotor system in both surgical and rehabilitative approaches. Current methods as leaflets or videos lacks of adherence control, evolution control and knowledge of how the patient do the exercises which compromise the expected results. Touch-screens of Tablet devices have showed a large potential to cover these needs and for the retraining of sensorimotor system. ReHand is a Tablet digital tool (Android and iOS) to prescribe and monitor exercise programs based on sensorimotor approach and developed under the guidelines of various healthcare professionals (hand surgeons, physiotherapists, rehabilitators and occupational therapists) to implement home exercise programs and monitor patients. Subjects are selected by emergency, hand surgery, rehabilitation and physiotherapy services of six hospitals from Andalusian Public Health Service through consecutive sampling. Concretely, patients over 18 years of age with trauma and soft injuries of the wrist, hand and fingers, no more than 10 days after surgery or removal of immobilization. Experimental group will receive access to ReHand app to perform a monitored home exercises program. Control group will receive the conventional method employed: a home exercise program in paper with recommendations. Clinical variables will be assessed at baseline before group allocation, 4 weeks, 3 months and 6 months. At the end of the study, cost-utility variables will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patients with trauma or soft tissue injuries of the wrist, hand and fingers. Dupuytren, carpal tunnel syndrome, rizarthrosis, distal radius fracture, carpal fracture or metacarpal fracture.

Exclusion Criteria:

* Neurological pathology that affects the upper limb.
* Non-cooperative.
* Psychiatric illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Self-reported functional ability using the validated Spanish version of the QuickDASH in patients with hand conditions. | Change from Baseline QuickDASH at one month, three months and six months.
  The shortened form of the DASH questionnaire (Disabilities of the Arm, Shoulder and Hand questionnaire) is an 11-item questionnaire that measures patient's ability to complete tasks, absorb forces, and severity of symptoms.
Wrist pain and disability in activities of daily living is assessed using the Spanish version of the 15-item questionnaire Patient Rated Wrist Evaluation (PRWE). | Change from baseline PRWE at one month, three months and six months.
  The PRWE comprises a 5-item pain subscale and a 10-item function subscale. The final score is between 0 - 100 points with higher scores indicating more disability.

SECONDARY OUTCOMES:
Dexterity assessed using the Nine Hole Peg Test | Change from baseline Nine Hole Peg Test at one month and three months.
  This test consists of placing nine small cylinders in the nine holes in the base or container of the "Nine Hole Peg Test".
Grip strength assessed using a hydraulic grip dynamometer | Change from baseline Grip strength at one month and three months.
  The Maximun power of the hand muscles used to firmly grasp an object by wrapping the fingers around it, pressing it against the palm, and using the thumb to apply counter-pressure, using a Hydraulic grip dynamometer.
Self-reported pain assessed using a Visual Analog Scale (VAS) of pain. | Change from baseline Visual Analog Scale of Pain at one month and three months.
  Participants report their pain intensity using the 0 to 10 VAS, where 0 refers to "no pain" and 10 refers to "the worst imaginable pain".
Joint position sense test | Change from baseline Joint position sense at one month and three months.
  A test to evaluate the ability to accurately reproduce a specific joint angle without the vision of the joint.
Quality of life is assessed using the Spanish version of the self-completion EQ-5D-5L questionnaire | Change from baseline EQ-5D-5L Questionnaire at one month and three months.
  Brief questionnaire which evaluated health state is in 5 domains: mobility, capacity for self-care, conduct of usual activities, pain or discomfort and anxiety or depression
Wrist flexion and extension range of movement. | Change from baseline wrist flexion and extension range of movement at one month and three months.
  Wrist flexion and extension range of movement assessed using a standard goniometer.
Economic factors relating to cost-utility. | Chage from baseline Economic factors relating to cost-utility at six months.
  Absence due to illness, use of health resources (number of consultations to specialist doctor, physiotherapy occupational therapy sessions, emergency department), time frame in rehabilitation services.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen de la Macarena, Seville, Andalusia
  - University of Seville, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suero-Pineda A, Oliva-Pascual-Vaca A, Duran MR, Sanchez-Laulhe PR, Garcia-Frasquet MA, Blanquero J. Effectiveness of a Telerehabilitation Evidence-Based Tablet App for Rehabilitation in Traumatic Bone and Soft Tissue Injuries of the Hand, Wrist, and Fingers. Arch Phys Med Rehabil. 2023 Jun;104(6):932-941. doi: 10.1016/j.apmr.2023.01.016. Epub 2023 Feb 8. PMID 36758713